CLINICAL TRIAL: NCT04085900
Title: Searching for Early Detection Biomarkers of Nasopharyngeal Carcinoma in Zhongshan City
Brief Title: Screening Nasopharyngeal Carcinoma With EBV Associated Biomarkers in Zhongshan City
Status: Recruiting | Type: Observational
Sponsor: Zhongshan People's Hospital, Guangdong, China (Other)
Collaborators: Wuzhou Red Cross Hospital (Other); Xiamen University (Other)
Responsible Party: Principal Investigator, Mingfang Ji, Dr. Mingfang Ji, Zhongshan People's Hospital, Guangdong, China
Other Study IDs: NPC-PRO-003
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Screening; Nasopharyngeal Carcinoma; Biomarker
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Blood Specimen Collection; Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood and saliva samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Screening cohort: 30-69 years old healthy participants in Zhongshan and Wuzhou.
  Interventions: Biological: Blood and saliva; Diagnostic Test: P85-Ab, EBNA1-IgA, VCA-IgA and EBV DNA; Diagnostic Test: Fiberoptic endoscopy and biopsy

INTERVENTIONS:
Biological: Blood and saliva — Collect blood and saliva samples from participants
Diagnostic Test: P85-Ab, EBNA1-IgA, VCA-IgA and EBV DNA — Detect P85-Ab, EBNA1-IgA, VCA-IgA for all participants, and detect EBV DNA for all male participants and P85-Ab positive female participants.
Diagnostic Test: Fiberoptic endoscopy and biopsy — Screening participants will refer to fiberoptic endoscopy and biospy

SUMMARY:
All participants will be tested for EBV associated biomarkers, including EBNA1-IgA, VCA-IgA, BNLF2b total antibodies (P85-Ab) et al. For all male participants and P85-Ab positive female participants, EBV DNA in plasma will be tested. Screening positive participants will be followed up annually.

All subjects will also be followed by record linkage to Cancer Register and Population Register.

DETAILED DESCRIPTION:
Sample selection

- Select communities of 20,000 to 40,000 populations in Zhongshan City and Wuzhou city as the investigators' fields.

Participants recruitment

* Subjects voluntarily attend this screening study Informed consent - Informed consent forms will be collected at the recruitment. Questionnaires.
* Face-to-face interviews are conducted by well-trained investigators.

Tests and follow up

* At initial screening, all participants will be tested for EBV associated biomarkers, including EBNA1-IgA, VCA-IgA, P85-Ab et al. And in males, EBV-DNA will be tested. Based on EBNA1-IgA, VCA-IgA, participants will be stratified into high, moderate and low risk. Screening positive include P85-Ab positive, high or moderate risk of NPC or EBV DNA positive. The rest will be screening negative.
* During the initial screening and following up, people with high risk or P85-Ab positive will refer to the diagnostic workup for NPC. Briefly, fiberoptic endoscopy and pathological biopsy will be performed by otorhinolaryngologists.
* Screening positive people not diagnosed as nasopharyngeal carcinoma in the first year will be followed up annually.
* EBV DNA single positive people will refer to the diagnostic workup for NPC in the third year of follow up.
* The rest of the blood samples will be stored at the biobank of Zhongshan People's Hospital for further research.
* All subjects will also be followed by record linkage to Cancer Register and Population Register.

ELIGIBILITY:
Inclusion Criteria:

* Subject residents in Zhongshan City or Wuzhou City
* Subject has no medical record of nasopharyngeal carcinoma
* ECOG 0-2
* Subject is able to comprehend, sign, and date the written informed consent document to participate in the study.
* Subject has psychical condition and well consciousness, and also accept and cooperate with the follow-up of this study.

Exclusion Criteria:

* Subject has heavy cardiovascular, liver or kidney disease.
* Subject has contraindications to nasopharyngeal fiberoptic endoscopy.

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30-69 years old healthy residences in Zhongshan City and Wuzhou City.
Sampling Method: Non-Probability Sample
Enrollment: 40000 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of different EBV associated biomarkers | 5 years
  To compare the sensitivity and specificity of different EBV associated biomarkers for NPC
Positive and negative predictive values of different EBV associated biomarkers | 5 years
  To compare the positive and negative predictive values of different EBV associated biomarkers for NPC

SECONDARY OUTCOMES:
Number needed to screen to identify one nasopharyngeal carcinoma | 5 years
  To compare the number of participants needed to screen identify one nasopharyngeal carcinoma for different biomarkers
Early diagnosis rate of nasopharyngeal carcinoma | 5 years
  To compare the early diagnosis rate of different biomarkers for nasopharyngeal carcinoma

OTHER OUTCOMES:
The health economic benefits of different biomarkers for nasopharyngeal carcinoma | 5 years
  To explore the overall survival rate, progression free survival rate and health economic benefits of NPC screening using different biomarkers
New screening strategy of nasopharyngeal carcinoma screening | 5 years
  Comprehensive analysis of the performance of different biomarkers and their combination in the screening of nasopharyngeal carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Mingfang Ji, MD, Principal Investigator — Zhongshan People's Hospital, Guangdong, China
Locations (2):
- China (2):
  - Zhongshan People's Hospital, Zhongshan, Guangdong
  - Wuzhou Red Cross Hospital, Wuzhou, Guangxi

REFERENCES:
- [Derived] Li T, Li F, Guo X, Hong C, Yu X, Wu B, Lian S, Song L, Tang J, Wen S, Gao K, Hao M, Cheng W, Su Y, Zhang S, Huang S, Fang M, Wang Y, Ng MH, Chen H, Luo W, Ge S, Zhang J, Xia N, Ji M. Anti-Epstein-Barr Virus BNLF2b for Mass Screening for Nasopharyngeal Cancer. N Engl J Med. 2023 Aug 31;389(9):808-819. doi: 10.1056/NEJMoa2301496. PMID 37646678